CLINICAL TRIAL: NCT00626067
Title: Pilot Study of Patient Acceptance and Impact of the New Travatan™ Compliance Monitoring Dispenser (Travatan™ Dosing Aid)
Brief Title: Study of Patient Use and Perception of the Travatan Dosing Aid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jonathon Myers, Attending Surgeon, Wills Eye
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB #06-762E; CMS-06-09 (Other: Wills Eye Hospital)
Record Dates: First submitted 2008-01-22; First posted 2008-02-29 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Glaucoma
Keywords: Travatan Dosing Aid; compliance monitoring dispenser
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Fully functional monitoring device (Active Comparator): Fully functional monitoring device
  Interventions: Device: Fully functional monitoring device
- 2 Partially functional monitoring device (Active Comparator): Partially functional monitoring device
  Interventions: Device: Partially functional monitoring device
- 3 Non-functional monitoring device (Sham Comparator): Non-functional monitoring device
  Interventions: Device: Non-functional monitoring device

INTERVENTIONS:
Device: Fully functional monitoring device — Pt received fully functional monitoring dispenser for use with their Travatan eye drops
  Arms: 1 Fully functional monitoring device
Device: Partially functional monitoring device — Patient received a particually functional Travatan Compliance Monitoring Dispenser
  Arms: 2 Partially functional monitoring device
Device: Non-functional monitoring device — Patient received a non functioning Travatan Compliance Monitoring Dispenser
  Arms: 3 Non-functional monitoring device

SUMMARY:
The primary objective of this study is to determine the opinions of patients who are given the Travatan Compliance Monitoring Dispenser to use to dispense their Travatan glaucoma drops.

DETAILED DESCRIPTION:
Patients enrolled in this study will use the new Travatan compliance monitoring dispenser for 6 weeks. Patients will be informed that some, but not all, patients' compliance will be monitored by the device. Patients are randomly assigned to one of three groups (proportionally in a 2/2/1 ratio):

1. Fully functional Travatan compliance monitor
2. Travatan compliance monitor with LCD display and alarms disabled, but compliance monitoring intact
3. Travatan compliance monitor with LCD display, alarms and compliance monitor disabled.

At end of study, patients fill out questionnaire assessing

1. Patient opinion regarding device: ease of use of new device; preference vs Travatan use without device, etc
2. patient's belief as to whether their compliance was monitored or not

Rates of adherence are compared across groups and with regard to patients' reported beliefs as to whether they were monitored.

The design of this study should allow the clinicians to ethically monitor compliance in patients who do and do not believe that they are being monitored. The use of monitoring devices without a functioning display and alarm should lead to some patients believing that they are not being monitored. As patients are told at the outset that they may or may not be monitored, this should be an ethically acceptable design. However, the collected data will allow a preliminary assessment of the impact of the patients' beliefs as to whether they are being monitored on their actual compliance, and hence an additional potential value of the device.

ELIGIBILITY:
Inclusion Criteria:

* Open angle glaucoma or ocular hypertension
* Presently using Travatan eye drops

Exclusion Criteria:

* Allergy to prostaglandin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Assess patients' opinions regarding new Travatan Compliance Monitoring Dispenser | 6 weeks

SECONDARY OUTCOMES:
Pilot study of the impact of physician monitoring of compliance on patient compliance | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Myers, MD, Principal Investigator — Wills Eye Institute

IPD SHARING:
Plan to Share IPD: Yes
A Manuscript has been accepted and published in Patient Preference and Adherence.

REFERENCES:
- See also: Patient Preference and Adherence — https://doi.org/10.2147/PPA.S114746